CLINICAL TRIAL: NCT05555524
Title: Effect of Cool Baby Oil on Pruritus and Sleep Quality Among Uremic Patients: a Double-blind Placebo-controlled Randomized Clinical Trial
Brief Title: Cool Baby Oil for Pruritus and Sleep Quality Among Uremic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Maha Gamal Ramadan Asal, Principle investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022-9-43
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Haemodialysis-Associated Pruritus

STUDY DESIGN:
Intervention Model Description: two-group pre-test and repeated post-test study
Who Masked: Participant, Outcomes Assessor
Masking Description: A two computer allocation sequence will be generated. They will be placed in an opaque, sealed envelope and kept with the head nurse of each hemodialysis unit. After completing the baseline data, the clinical researchers open the envelops and assign the patients to one group. The baby oil and the placebo distilled water will be placed on identical bottles and participants will not be informed about group assignments. The clinical researcher will label the groups as A or B; only the clinical researchers will know the group allocation. Both the outcome assessor and the statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baby oil (Experimental): A cool commercial baby oil at a temperature between 10°C and 15°C that composed of Paraffinum Liquidum, Isopropyl Palmitate, Parfumwill be applied to the affected area for a period of 15-20 min for three times a week before each hemodialysis session for 12 weeks.
  the baby oil bottle will be stored at the refrigerator.
  Interventions: Other: Baby oil
- Placebo (Placebo Comparator): A cool distilled water at a temperature between 10°C and 15°C with added two drops of the baby oil to each 100 cc will be applied to the affected area for a period of 15-20 min for three times a week before each hemodialysis session for 12 weeks.
  the distilled water will be put at an identical bottle as the baby oil bottle and stored at the refrigerator.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Baby oil — Before each application
  * Hand hygiene will be done
  * Skin care will be done to the affected area and the area is thoroughly dried.
  * Participants will wear a hospital gown and seated comfortably on their bed.
  * Gentle massage with the cool baby oil will be applied on the itching area and is continued for 15-20 min.
  * Message will be applied for three times a week before each hemodialysis session for 12 weeks
  Arms: Baby oil
Other: Placebo — Before each application
  * Hand hygiene will be done
  * Skin care will be done to the affected area and the area is thoroughly dried.
  * Participants will wear a hospital gown and seated comfortably on their bed.
  * Gentle massage with the cool distilled water will be applied on the itching area and is continued for 15-20 min.
  * Message will be applied for three times a week before each hemodialysis session for 12 weeks
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effect of cool baby oil on pruritus and sleep quality among uremic patient

Research Hypothesis:

* H01: There is no difference between hemodialysis patients with uremic pruritus who apply cool baby and those who apply placebo regarding sleep quality at 4 weeks follow-up
* H02: There is no difference between hemodialysis patients with uremic pruritus who apply cool baby and those who apply placebo regarding itching severity at 4 weeks follow-up
* H03: There is no difference between hemodialysis patients with uremic pruritus who apply cool baby and those who apply placebo regarding sleep quality at 12 weeks follow up
* H04: There is no difference between hemodialysis patients with uremic pruritus who apply cool baby and those who apply placebo regarding itching severity at 12 weeks follow up
* H1: Hemodialysis patients with uremic pruritus who apply cool baby oil will exhibit improved sleep quality than those who apply placebo at 4 weeks follow up
* H2: Hemodialysis patients with uremic pruritus who apply cool baby oil will exhibit decreased itching severity than those who apply placebo at 4 weeks follow up
* H3: Hemodialysis patients with uremic pruritus who apply cool baby oil will exhibit improved sleep quality than those who apply placebo at 12 weeks follow up
* H4: Hemodialysis patients with uremic pruritus who apply cool baby oil will exhibit decreased itching severity than those who apply placebo at 12 weeks follow up

DETAILED DESCRIPTION:
Treatment of uremic pruritus is difficult due to the refractory nature of the disease, resulting in poor hemodialysis patient quality of life, pharmacological therapy is the most common clinical treatment method. Unfortunately, despite these interventions, pruritus remains a chronic problem for many dialysis patients. Recently, non-pharmacological interventions are effective for hemodialysis patients with uremic pruritus. Emollients that include Petrolatum, lanolin, mineral oil, and dimethicone were very effective, readily available, and cost-effective interventions in comparison to other methods to improve pruritus symptoms. Several studies have been conducted and show the efficiency of baby oil in controlling pruritus and enhancing sleep quality among hemodialysis patients. However these studies evaluate the short-term effect (4 weeks), Although these studies employed usual care, no-treatment group as the control condition, thus it was not possible to blind the participants. This type of control group would likely increase treatment effects from baby oil by comparison. Thus the current study will be conducted to evaluate the effect of baby oil on pruritus and sleep quality compared to a placebo control at 4 and 12 weeks followup.

ELIGIBILITY:
Inclusion Criteria:

* Having three episodes of itching (each episode 5 min or longer) within the last 2 weeks
* Having intermittent itching complaints during the last 6 month
* Agreed to be on a fixed dose of the medical treatment throughout the study

Exclusion Criteria:

* Open wound
* Skin infection
* Edema
* History of allergic reaction to the oils
* Liver and dermatological diseases
* Usage of other treatment rather than the medical treatment on a regular basis 2 weeks prior to randomization and throughout the study
* Currently participating in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-10-02 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
mean itching severity score at the baseline defined by Itching Severity Scale (ISS) | at the baseline (before assigning the participants to the study groups)
  this scale includes three items; (1) distribution of itching; (2) severity of itching; and (3) sleep disturbance caused by itching. Scores range 2-45. Increasing scores indicate increasing severity and intensity of itching.
change of the mean Itching Severity Scale (ISS) at 4 weeks | after 4 weeks from the baseline
  this scale includes three items; (1) distribution of itching; (2) severity of itching; and (3) sleep disturbance caused by itching. Scores range 2-45. Increasing scores indicate increasing severity and intensity of itching.
Change of the mean Itching Severity Scale (ISS) at 12 weeks | after 12 weeks from the baseline
  this scale includes three items; (1) distribution of itching; (2) severity of itching; and (3) sleep disturbance caused by itching. Scores range 2-45. Increasing scores indicate increasing severity and intensity of itching.
Mean pruritus severity Score on Visual Analog Scale at the Baseline | at the baseline (before assigning the participants to the study groups)
  This scale will be used to measure the itching intensity and consisting of a 10cm long line and a single question. The left end point represents "no itch" and the right end point the "worst imaginable itch
Change from baseline mean of the pruritus severity score on the Visual Analog Scale at 4 weeks | after 4 weeks from the baseline
  This scale will be used to measure the itching intensity and consisting of a 10cm long line and a single question. The left end point represents "no itch" and the right end point the "worst imaginable itch
Change from baseline mean of the pruritus scores on the Visual Analog Scale at 12 weeks | after 12 weeks from the baseline
  This scale will be used to measure the itching intensity and consisting of a 10cm long line and a single question. The left end point represents "no itch" and the right end point the "worst imaginable itch
Mean score of the sleep quality on the Pittsburgh sleep quality index at the baseline | at the baseline (before assigning the participants to the study groups)
  it measure the self-rated sleep quality over the past month, and it is consisted of 19 self-rated question and 5 question rated by bed partner or roommate. Score ranges from 0 to 21.
  a score of > 5 indicate poor or difficult sleep and a score of ≤ 5 indicate good-sleep .
Change from baseline mean of the sleep quality on the Pittsburgh sleep quality index at 4 weeks | after 4 weeks from the baseline
  it measure the self-rated sleep quality over the past month, and it is consisted of 19 self-rated question and 5 question rated by bed partner or roommate. Score ranges from 0 to 21.
  a score of > 5 indicate poor or difficult sleep and a score of ≤ 5 indicate good-sleep .
Change from baseline mean of the sleep quality on the Pittsburgh sleep quality index at 12 weeks | after 12 weeks from the baseline
  it measure the self-rated sleep quality over the past month, and it is consisted of 19 self-rated question and 5 question rated by bed partner or roommate. Score ranges from 0 to 21.
  a score of > 5 indicate poor or difficult sleep and a score of ≤ 5 indicate good-sleep .

SECONDARY OUTCOMES:
socio-demographic and clinical data assessment tool | (before assigning the participants to the study groups)
  this tool gathers data about participants' age, gender, educational level, marital status, area of residence, and occupation, duration of disease, comorbidity disease, duration of itching, Concurrent use of antihistamine for itching, period of most intense pruritus.
Related adverse Events | from starting of the intervention till 2 days after study completion
  An unfavorable change in the health of a participants that happens during a clinical study or within a 2 days after the study has ended. This change may or may not be caused by the assigned treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Maha G Asal, Phd, Principal Investigator — Alexandria University; Hoda A El-Deeb, Phd, Principal Investigator — Alexandria University; Mona A Amer, Phd, Principal Investigator — Alexandria University; Mervat A Hawash, Phd, Principal Investigator — Alexandria University
Locations (2):
- Egypt (2):
  - Dialysis Units of Almowasah University Hospital, Alexandria
  - Dialysis Units of the Main University Hospital, Alexandria

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make individual participant data available.